CLINICAL TRIAL: NCT04350450
Title: Hydroxychloroquine Treatment of Healthcare Workers With COVID19 Illness at Montefiore: a Review of Process Feasibility, Safety, and Clinical Outcomes
Brief Title: Hydroxychloroquine Treatment of Healthcare Workers With COVID19 Illness at Montefiore
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI withdrew the submission to the IRB
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Priya Nori, Principal Investigator, Montefiore Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-11445
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-04

CONDITIONS: COVID; Coronavirus; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): Eligible participants will be offered the standard Montefiore HCQ dosing regimen of 400mg every 12 hours x 24 hours, then 400mg daily for remaining 4 days and complete a survey study
  Interventions: Drug: Hydroxychloroquine
- Control Group (No Intervention): Participants who opt not to receive the study drug will also be invited to participate in the survey study assessing COVID19 symptoms

INTERVENTIONS:
Drug: Hydroxychloroquine — 400 mg tablet
  Arms: Treatment Group

SUMMARY:
Given the high prevalence of COVID19 illness (both SARS-CoV-2 RT-PCR confirmed and highly suspect cases) among healthcare workers (HCW) within the Montefiore Health System (MHS), hydroxychloroquine (HCQ) will be prescribed to healthcare workers who are at the highest risk for severe COVID19 illness.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic with COVID illness (either RT-PCR test confirmed or highly suspect clinical symptoms)
* Call into office within the first 7 days of illness
* Have any of the following high risk conditions:

  * Age >60
  * HTN, CAD, or chronic heart disease
  * Diabetes
  * Chronic kidney disease
  * Chronic lung disease
  * Active or recent chemotherapy for malignancy
  * Organ transplant
  * Taking Immune-suppressing medications
  * HIV with CD4 <200 cells/mm3
* Experiencing at least one of the following high risk symptoms:

  * Severe cough
  * Fever 100.0F or greater
  * Diarrhea
  * Shortness of Breath
  * Hypoxia

Exclusion Criteria:

• HCW not meeting high-risk criteria or those with a contraindication to HCQ will not be offered HCQ

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Time to resolution of symptoms | up to 4 weeks
  Time that it takes for symptoms to be resolved in those who were treated vs untreated

SECONDARY OUTCOMES:
Number of days from onset of illness to symptom resolution | up to 4 weeks
Number of days to return to work | up to 4 weeks
Rate of hospital admission in treated and untreated healthcare workers | up to 4 weeks
Adverse effect of HCQ during treatment | up to 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Priya Nori, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No